CLINICAL TRIAL: NCT06503549
Title: Investigation of Tactile Acuity, Right-left Discrimination, and Motor Imagery in Chronic Rotator Cuff-related Shoulder Pain - A Case Control Study
Brief Title: Tactile Acuity, Right-left Discrimination, and Motor Imagery in Chronic Rotator Cuff-related Shoulder Pain
Status: Completed | Type: Observational
Sponsor: Acibadem University (Other)
Responsible Party: Principal Investigator, Nuray Alaca, Prof Dr., Acibadem University
Other Study IDs: 2023/32-18
Record Dates: First submitted 2024-07-10; First posted 2024-07-16 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Shoulder Pain; Rotator Cuff Syndrome
MeSH Terms: conditions — Shoulder Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy control
  Interventions: Other: Assessments
- Patient with rotator cuff-related shoulder pain
  Interventions: Other: Assessments

INTERVENTIONS:
Other: Assessments — Only the current assessments will be made

SUMMARY:
A common finding in various chronic musculoskeletal pain conditions is changes in the cortical sensorimotor region. Functional brain changes associated with chronic pain include changes in the working body schema and associated mechanisms. However, the number of studies on this subject is quite limited, especially in the shoulder joint. There is no study on rotator cuff-related shoulder pain. In the light of this information, the present study aims to compare tactile acuity, right-left reasoning ability and motor imagery ability in chronic rotator cuff-related shoulder pain with healthy controls. In addition, the relationship of these markers with pain level, pressure pain threshold, range of motion, functionality, pain-related fear and central synthesis level will be investigated as a secondary objective.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years
* Participants were classified with chronic Chronic Rotator Cuff-related Shoulder Pain if duration was equal or greater than 6 months, as recommended by the International Association for the Study of Pain for research purposes
* Pain at rest maximum 2 out of 10 on verbal numerical rating scale
* Pain over the deltoid and/or upper arm region for more than 4 weeks, pain associated with arm movement, and familiar pain reproduced with loading or resisted testing during abduction or external rotation of the arm
* Patient had to test positive at least 3 out of 5 symptoms-provoking tests: pain during Neer test, Hawkins-Kennedy test, Jobe test, painful arc between 60° and 120°, pain or weakness during external rotation resistance test

Exclusion Criteria:

* Bilateral shoulder pain
* Corticosteroid injections less than 6 weeks prior to the enrolment
* Participants who were pregnant, Mini Mental State Examination score >24
* Clinical signs of full-thickness rotator cuff tears (positive external and internal rotation lag tests or drop arm test)
* Evidence of adhesive capsulitis (50% or more than 30° loss of passive external rotation)
* Previous cervical, thoracic or shoulder surgery; recent fractures or dislocations on the painful shoulder
* Symptoms of cervical radiculopathy as primary complaint (tingling, radiating pain in the arm associated with neck complaints)
* Primary diagnosis of acromioclavicular pathology, shoulder instability
* Previous medical imaging confirming full-thickness rotator cuff tears or calcifications larger than 5mm
* Patients with competing pathologies (inflammatory arthritis, neurological disorders, fibromyalgia, malignancy)
* History of cancer, neurologic, systemic, rheumatic or vascular disorder and use of psychiatric medication
* Participants performing overhead sport activities for more than 4hours/week

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 18 and 65 years old were eligible to participate if they had rotator cuff related shoulder pain
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-07-15 (Actual); Study Completion 2024-08-06 (Actual)

PRIMARY OUTCOMES:
Tactile Acuity (The two-point discrimination test) | Baseline
  The two-point discrimination test is used to assess if the patient is able to identify two close points on a small area of skin, and how fine the ability to discriminate this are. It is a measure of tactile agnosia, or the inability to recognize these two points despite intact cutaneous sensation and proprioception
Left/right discrimination (Lateralization) | Baseline
  Right-Left Discrimination will be evaluated with Recognise™ applications (Shoulder and Hand) developed by the "Neuro Orthopedic Institute".
Kinesthetic and Visual Imagery Questionnaire (KVIQ) | Baseline
  Motor imagery ability will be assessed with the Kinesthetic and Visual Imagery Questionnaire (KVIQ). The participant gives a score between 1 and 5 for the image he/she imagines: "1 point: no image, 5 points: as clear as the original." This process is repeated for each task and at the end of the survey, kinesthetic imagery score, visual imagery score and total score are calculated.
Pressure Pain Threshold | Baseline
  A digital pressure algometer will be applied to the web space of the foot opposite the trigger point. Participants are instructed to say "stop" or "pain" so the stimulus can be terminated "when the sensation first transitions from pressure to pain" (pain threshold).
Central Sensitization Scale | Baseline
  Central Sensitization Scale, which can be applied in the presence of chronic pain, is used in central sensitization syndromes. It consists of two parts. Part A of the scale includes a Likert scale (0-4 points) that questions health-related symptoms. This section is scored from 0 to 100, with higher numbers being associated with a higher degree of central sensitization. Scores of 40 and above indicate the presence of central sensitization. In section B, it questions whether any of the central sensitization syndromes have been diagnosed before.

SECONDARY OUTCOMES:
The Numerical Rating Scale (NPRS-11) | Baseline
  the Numerical Rating Scale (NPRS-11) is an 11-point scale for self-report of pain. It is the most commonly used unidimensional pain scale. The respondent selects a whole number (integers 0-10) that best reflects the intensity (or other quality if requested of his/her pain).0 point is the minimum and 10 point is the maximum. The higher the score, the more severe the pain.
The Shoulder Pain and Disability Index | Baseline
  The Shoulder Pain and Disability Index (SPADI) was developed to measure current shoulder pain and disability in an outpatient setting. The SPADI contains 13 items that assess two domains; a 5-item subscale that measures pain and an 8-item subscale that measures disability between 0 to 100, with a higher value indicating worse condition.
Shoulder mobility on the Shoulder Range of Motion | Baseline
  Shoulder ROM was measured in six directions (Flexion, Extension, Abduction, Adduction, Right rotation, Left rotation, degree) with goniometer.
Pain Catastrophizing Scale | Baseline
  The Pain Catastrophizing Scale (PCS) is a 13-item self-report measure designed to assess catastrophic thinking related to pain among adults with or without chronic pain.The person may score a total of 52 (Pain Catastrophizing Scale). A high score indicates a high level of catastrophic.
Fear avoidance belief questionnaire (FABQ) | Baseline
  Fear avoidance belief questionnaire FABQ) is a questionnaire based on the fear-avoidance model of exaggerated pain perception. The FABQ measures patient's fear of pain and consequent avoidance of physical activity (PA) because of their fear.There is a maximum score of 96. A higher score indicates more strongly held fear avoidance beliefs. There are two subscales within the FABQ; the work subscale (FABQw) with 7 questions (maximum score of 42) and the physical activity subscale (FABQpa) with 4 questions (maximum score of 24)

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Acıbadem University, Istanbul
  - Dokuz Eylül University, Izmir

IPD SHARING:
Plan to Share IPD: Undecided